CLINICAL TRIAL: NCT06669429
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effects of RS-C1001 Tablets in Chinese Healthy Subjects
Brief Title: A Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RS-C1001 Tablets in Chinese Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Director of the Institute of Clinical Pharmacology, Peking University First Hospital, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RS-C1001-C-1-1-001
Record Dates: First submitted 2024-10-12; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Dyslipidemia
Keywords: RS-C1001 tablets Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Part A1-RS-C1001 tablet dose 1 (Experimental)
  Interventions: Drug: RS-C1001
- Cohort 2: Part A1-RS-C1001 tablet dose 2/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 3: Part A1-RS-C1001 tablet dose 3/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 4: Part A1-RS-C1001 tablet dose 4/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 5: Part A1-RS-C1001 tablet dose 5/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 6: Part A1-RS-C1001 tablet dose 6/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 7: Part A1-RS-C1001 tablet dose 6/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 8: Part A1-RS-C1001 tablet dose 8/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 9: Part A1-RS-C1001 tablet dose 9/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: placebo
- Cohort 10: Part A1-RS-C1001 tablet dose 10/placebo tablet (Experimental)
  Interventions: Drug: RS-C1001; Drug: Placebo

INTERVENTIONS:
Drug: RS-C1001 — Subjects will receive RS-C1001 tablets orally as a single ascending dose
  Arms: Cohort 1: Part A1-RS-C1001 tablet dose 1; Cohort 2: Part A1-RS-C1001 tablet dose 2/placebo tablet; Cohort 3: Part A1-RS-C1001 tablet dose 3/placebo tablet; Cohort 4: Part A1-RS-C1001 tablet dose 4/placebo tablet; Cohort 5: Part A1-RS-C1001 tablet dose 5/placebo tablet; Cohort 6: Part A1-RS-C1001 tablet dose 6/placebo tablet
Drug: RS-C1001 — Subjects will receive RS-C1001 tablets orally as a multiple ascending dose
  Arms: Cohort 7: Part A1-RS-C1001 tablet dose 6/placebo tablet; Cohort 8: Part A1-RS-C1001 tablet dose 8/placebo tablet; Cohort 9: Part A1-RS-C1001 tablet dose 9/placebo tablet
Drug: RS-C1001 — Subjects will receive RS-C1001 tablets orally as a single dose after intake of a high-calorie, high-fat breakfast
  Arms: Cohort 10: Part A1-RS-C1001 tablet dose 10/placebo tablet
Drug: placebo — Subjects will receive placebo matching tne RS-C1001 dose orally as a single ascending dose
  Arms: Cohort 2: Part A1-RS-C1001 tablet dose 2/placebo tablet; Cohort 3: Part A1-RS-C1001 tablet dose 3/placebo tablet; Cohort 4: Part A1-RS-C1001 tablet dose 4/placebo tablet; Cohort 5: Part A1-RS-C1001 tablet dose 5/placebo tablet; Cohort 6: Part A1-RS-C1001 tablet dose 6/placebo tablet
Drug: placebo — Subjects will receive placebo matching tne RS-C1001 dose orally as a multiple ascending dose
  Arms: Cohort 7: Part A1-RS-C1001 tablet dose 6/placebo tablet; Cohort 8: Part A1-RS-C1001 tablet dose 8/placebo tablet; Cohort 9: Part A1-RS-C1001 tablet dose 9/placebo tablet
Drug: Placebo — Subjects will receive placebo matching tne RS-C1001 dose orally as a single dose after intake of a high-calorie, high-fat breakfast
  Arms: Cohort 10: Part A1-RS-C1001 tablet dose 10/placebo tablet

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food effects of RS-C1001 tablets in Chinese healthy subjects.

This study will consist of two parts (Parts A and B). 42 subjects have been planned for Part A and 30 subjects for Part B.

DETAILED DESCRIPTION:
This is a Phase I, First In Human (FIH), randomized, double-blind, placebo-controlled study in Chinese healthy subjects.

42 subjects have been planned for Part A and 30 subjects for Part B.

Part A:

A Screening Period of maximum 14 days. Admission to study center (Day -1). A Treatment Period (Day 1 to Day 4) with a single dose of RS-C1001 or placebo on Day 1. Subjects will be discharged on Day 4.

A Follow-up Visit within 6 to 8 days after the Investigational Medicinal Product (IMP) dose for all cohorts.

(i) Part A1 - Up to 6 dose cohorts of RS-C1001 are planned to be investigated. Two subjects (one male and one female) planned to be enrolled in the 50 mg dose cohort will receive the investigational drug orally. The remaining 5 dose cohorts, 6 subjects will be randomized to receive RS-C1001, and 2 subjects randomized to receive placebo.

(ii) Part A2 - The subjects from a chosen cohort in Part A1 will return to the study center no sooner than 7 days after the first dose administration of IMP and will receive RS-C1001 or placebo after intake of a high-calorie, high-fat breakfast, to assess the effect of food on the PK of RS-C1001.

The subjects will stay at the study center until 72 hours post-dose in both the parts.

• Part B: Multiple Ascending Dose (MAD) cohort - Up to 3 dose cohorts are planned to be investigated. In each cohort, 10 subjects will participate and receive either RS-C1001 or placebo, randomized 4:1 for 10 days dosing.

Subjects will be discharged on Day 13. A Follow-up Visit within 15 to 17 days after the Investigational Medicinal Product (IMP) dose for all cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should fully understand the purpose, nature, method and possible adverse reactions of the test, and voluntarily sign the informed consent.
2. Healthy subjects aged 18-45 years old (including boundary values, subject to the time of signing the informed consent form), regardless of gender;
3. Have a BMI between 19 and 26 kg/m2 (including the boundary value), and the weight of males is not less than 50 kg, and the weight of females is not less than 45 kg;
4. Researchers determine that the overall health status of the subjects is good based on their medical history, physical examination, vital signs, 12 lead electrocardiogram , laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function, early kidney damage detection), virus serology, and other results (normal or abnormal examination results have no clinical significance);
5. The serum LDL-C of the enrolled subjects in MAD study is less than 4.1 mmol/L, and the serum TG is less than 3.4 mmol/L.
6. Female participants must be in a negative pregnant and non lactating state; And female subjects of childbearing age and male subjects with female partners of childbearing age agree to use contraception from the screening period until 6 months after the last dose (using medically recognized effective contraceptive measures). Male subjects can only donate sperm 6 months after the last dose.

Exclusion Criteria:

1. Individuals with a history of drug or other allergies, or those who may be allergic to the investigational drug or any component of the investigational drug as determined by the researcher;
2. Subjects with abnormal clinical manifestations, including but not limited to neurological, cardiovascular, blood, liver, kidney, gastrointestinal, respiratory, metabolic, endocrine, immune, and skeletal system diseases, who have been evaluated by the researchers as unsuitable for participation in this study;
3. Screening and baseline 12 lead electrocardiogram results (adjusted by Fridericia formula, QTcF=QT/(RR ^ 0.33), where RR=60/heart rate) for male subjects with QTcF (average of 3 consecutive test results) ≥ 450 ms and female subjects with QTcF ≥ 470 ms;
4. Subjects with eGFR<80 mL/min/1.73m ²;
5. Individuals who have a history of drug abuse within the past five years or have used drugs in the three months prior to screening, or who tested positive for drug abuse during screening or baseline;
6. Individuals who have smoked more than 5 cigarettes per day or habitually used nicotine containing products within the previous 3 months, or who are unable to quit smoking during the trial period;
7. Individuals who have consumed more than 14 units of alcohol per week within the previous 3 months (1 unit of alcohol=360 mL of beer, 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine), or have taken alcoholic products within 48 hours prior to receiving the test drug, or have tested positive for alcohol breath test at baseline;
8. Those who have suffered from clinically significant major diseases or undergone major surgical procedures within 28 days prior to receiving the investigational drug, or who are expected to undergo major surgery during the trial period;
9. If the researcher determines that any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health supplements have been used within 14 days before receiving the investigational drug, and the time interval between the start of the drug administration and the start of the trial is greater than 5 half lives, the corresponding subjects can also be enrolled; Within 30 days before accepting the investigational drug, use any known Chinese herbal medicine, vitamin, or tonic that can affect glucose and lipid metabolism (such as fish oil>1000 mg/day, drugs or health supplements containing Monascus rice ingredients);
10. Those who consume any food or beverage containing or metabolized to produce caffeine or xanthine (such as coffee, tea, chocolate) within 48 hours prior to receiving the investigational drug;
11. Screening period virus serological testing for subjects who are positive for human immunodeficiency virus antibodies (HIV Ab), HBV surface antigen (HBsAg), HCV antibodies (HCV Ab), or Treponema pallidum antibodies (TP Ab);
12. Those who have difficulty in venous blood collection or have a history of needle and blood dizziness;
13. Subjects with a history of grade 3 hypoglycemia;
14. Subjects who have used other clinical trial drugs or participated in clinical trials of medical devices within the past 3 months prior to receiving the investigational drug;
15. Subjects who have a history of blood donation or have lost more than 400 mL of blood in the three months prior to screening, or who plan to donate blood during the trial period;
16. The researcher believes that the participant is not suitable to participate in the trial due to other reasons or withdraws from the trial due to personal reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with Adverse Events (AEs) or Serious Adverse Events(SAEs). | Part A1 (SAD): Day1-7; Part A2 (FE): Day1-14; Part B (MAD): Day1-16
  Incidence, type, severity, and relationship of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 after single and multiple oral administration of RS-C1001 tablets in healthy male and female participants.
Numbers of participants with clinical laboratory tests abnormalities | Part A1 (SAD): Day2、Day4、Day7; Part A2 (FE): Day2、Day4、Day7、Day9、Day11、Day14; Part B (MAD): Day3、Day7、Day11、Day13、Day16
  Safety blood and urine samples collected are assessed for lab values that move out of the normal range will be noted and assessed for clinical significance. Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Numbers of participants with vital sign abnormalities | Part A1 (SAD): Day1-4、Day7; Part A2 (FE): Day1-4、Day7-11、Day14; Part B (MAD): Day1-13、Day16
  Numbers of participants with vital sign abnormalities
Numbers of participants with physical examination abnormalities | Part A1 (SAD): Day2、Day4、Day7; Part A2 (FE): Day2、Day4、Day7、Day9、Day11、Day14; Part B (MAD): Day3、Day7、Day11、Day13、Day16
  Numbers of participants with physical examination abnormalities
Number of participants with 12-lead electrocardiogram(ECG) abnormalities | Part A1 (SAD): Day1-4、Day7; Part A2 (FE): Day1-4、Day7-11、Day14; Part B (MAD): Day1-13、Day16
  Number of participants with 12-lead ECG abnormalities including PR, RR, QRS, QT and QTcF.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China